CLINICAL TRIAL: NCT04073641
Title: Danish Diabetes Barometer Survey 2019
Brief Title: Survey of People With Diabetes, Caregivers of People With Diabetes Parents of Children and Young People With Diabetes
Acronym: DiaBar2019
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: The Danish Diabetes Association (Other)
Responsible Party: Principal Investigator, Niels Ejskjær, Professor, Aalborg University Hospital
Other Study IDs: DiaBar2019
Record Dates: First submitted 2019-04-16; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey population: Adults with type 1 and type 2 diabetes and caregivers of people with diabetes including parents of children and young people with diabetes.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A survey of people with diabetes and caregivers of people with diabetes and parents of children and young people with diabetes in Denmark in order to assess perceived diabetes related health and wellbeing and perceived access to and gaps in medical care, support and other financial and support services.

DETAILED DESCRIPTION:
A questionnaire survey was designed for online completion by people with diabetes and caregivers of people with diabetes and parents of children and young people with diabetes in Denmark in order to assess their perceived diabetes related health and wellbeing and perceived access to and gaps in medical care, support and other financial and support services. The aim is for the survey to provide a cross-sectional assessment of present access to health, wellbeing and care for people with diabetes and caregivers in Denmark and to establish a survey tool suitable for ongoing long-term monitoring of well-being, care and support to people with diabetes and caregivers in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18

Exclusion Criteria:

* Not able to complete online questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with type 1 and type 2 diabetes, caregivers of people with diabetes and parents of children and young people with diabetes. Primary survey population are members of the national diabetes association.
Sampling Method: Non-Probability Sample
Enrollment: 10500 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-04-29 (Actual)

PRIMARY OUTCOMES:
Diabetes membership survey of health, access to care, support and services | The survey was administered from April 11 to 29th 2019
  Study-specific Likert-scale single item variables for perceived health, access to diabetes care, support and services (1-5)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Ejskjaer, PhD, Principal Investigator — Aalborg University Hospital; Soren E Skovlund, MSc, Study Director — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided